CLINICAL TRIAL: NCT01946555
Title: Prospective Longitudinal Observational Study to Evaluate the Clinical Characteristics and Opioids Treatments in Patients With Breakthrough Cancer Pain
Acronym: RER
Status: Completed | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: Studio RER
Record Dates: First submitted 2013-09-10; First posted 2013-09-19 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Tumor; Cancer Pain; Breakthrough Cancer Pain; Neuropathic Pain
Keywords: Breakthrough cancer pain; Neuropathic pain; Major opioid; Analgesics
MeSH Terms: conditions — Neoplasms; Cancer Pain; Neuralgia | interventions — Morphine; Fentanyl; Methadone; Buprenorphine; Oxycodone; Hydromorphone; Tapentadol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Worst pain, Average pain: It is necessary that patients are treated for their baseline pain with opioid medications 3rd step (WHO guidelines), having seven different provisions molecules (morphine, methadone, fentanyl, buprenorphine, oxycodone, hydromorphone and tapentadol), and that they receive opioid rescue medication, based on free choice among the options available on the market (in the form of transmucosal fentanyl: OTFC - lollipop, buccal buccal tablets, sublingual tablets, nasal spray in aqueous solution, with pectin nasal spray, morphine or other opioid "oral immediate release" or intravenously).
  Interventions: Drug: Morphine; Drug: Fentanyl; Drug: Methadone; Drug: Buprenorphine; Drug: Oxycodone; Drug: Hydromorphone; Drug: Tapentadol

INTERVENTIONS:
Drug: Morphine
Drug: Fentanyl
Drug: Methadone
Drug: Buprenorphine
Drug: Oxycodone
Drug: Hydromorphone
Drug: Tapentadol

SUMMARY:
The BTP (Breakthrough pain)was defined as "a transient exacerbation of pain that occurs either spontaneously, or in relation to a specific predictable or unpredictable trigger, despite relatively stable and adequately controlled background pain".

The BTP is a common clinical features in patients with cancer pain (BTcP: breakthrough cancer pain). The prevalence of BTcP is equal to 56%.

Currently, the investigators tend to recognize the idiopathic/spontaneous or accident BTcP in the three sub-types: voluntary, non- voluntary and procedural.

The diagnosis of BTCP is not always easy because in the cancer patient is normal to observe changes in the intensity of pain during the day, so it is necessary to differentiate slight fluctuations from the presence of real episodes of BTCP, for which is necessary to use a rescue treatment adjusted. In the study will be proposed the use of a diagnostic algorithm, present in the literature, to perform the diagnosis of BTCP.

In the presence of BTCP, is important both a correct controlled background pain with major opioids, which can reduce the number and the intensity of the painful episodes, both implement an adjunctive therapy, called "rescue", to be administered at the time which takes over the painful episode using, in this case, an opioid greater.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis (histologic or cytologic) of locally advanced cancer and / or metastatic disease;
* presence of baseline pain of moderate intensity / severe, necessitating treatment with opioids of the 3rd step / WHO, already in progress or to be undertaken at a stage just prior to the start of the study (see also criterion 4 where indicates that "the pain of base must be adequately controlled with opioids of the wHO 3rd step");
* estimated life expectancy of more than one month;
* presence of BTCP, diagnosed according to the criteria set by the definition of BTCP and the algorithm of Davies, for which it is established to undertake a treatment "rescue" of painful episodes, with the appropriate opioid drugs at the time of commencement of the study;
* capable of taking opioid medications for pain basic and breakthrough pain, by any route of administration;
* aged more than 18 years.

Exclusion Criteria:

* participation in other research projects that are in conflict or could confound the results of the study;
* absence of informed consent, or withdrawal of consent for study participation;
* presence of some pathological mental or psychiatric conditions, due to the tumor or concomitant diseases, which interfere with the state of consciousness or the ability to judge the point of jeopardizing the study protocol;
* need treatment for comorbid conditions present at the beginning of the study that could create potentially dangerous drug interactions with opioids (conazolici use of antifungals or macrolide antibiotics);
* contraindications of any kind for use of opioid drugs;
* positivity of a story, past or current, of substance abuse;
* inability to ensure regular follow-up;
* diagnosis of primary tumor of the brain;
* situation of the presence of BTCP already in treatment with opioid rescue of 3rd step;
* decision to use drugs "rescue" of different opioid 3rd step / WHO (NSAIDs, opioids of 2 ° step), for the treatment of BTCP;
* diagnosis of chronic renal failure proclaimed already in place, with values of blood creatinine ≥ 2 mg / dL.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study involves a longitudinal evaluation of BTCP in cancer patients with pain, through a follow-up of 4 weeks, which will examine in a dynamic clinical aspects (variation over time of the number and duration of episodes, painful intensity, changes in ATC and rescue therapy).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number and duration of episodes of BTcP | 28 days
Time to reach the peak of pain in the BTcP | 28 days
Maximum intensity of BTcP | 28 days

SECONDARY OUTCOMES:
Intensity of pain | 28 days
  Evaluate the relationship between the intensity of baseline pain in its various dimensions (worst, average and light on the last 24 hours) and intensity of pain reported during episodes of BTCP;
Effect of the treatments | 28 days
  Evaluate over time the effect of the treatments on the rescue BTCP, in terms of reduction of the number that the intensity of the episodes of BTCP

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Corli, MD, Principal Investigator — Mario Negri Institute of Pharmacological Research - IRCCS
Locations (11):
- Italy (11):
  - AO Universitaria Policlinico di Modena, Modena, Italia
  - A.O. Universitaria Parma, Parma, Italia
  - Ospedale Magati, Scandiano, Italia
  - Azienda USL - Ospedale di Carpi e Mirandola, Carpi
  - A.O.U. Arcispedale S. Anna, Ferrara
  - Ospedale di Fiorenzuola D'Arda, Fiorenzuola d'Arda
  - Ospedale di Lugo, Lugo
  - IRCCS-IRST Forlì, Meldola
  - Ospedale di Piacenza, Piacenza
  - Arcispedale S. Maria Nuova Azienda Ospedaliera, Reggio Emilia
  - Ospedale degli Infermi, Rimini

REFERENCES:
- [Background] Portenoy RK, Hagen NA. Breakthrough pain: definition and management. Oncology (Williston Park). 1989 Aug;3(8 Suppl):25-9. PMID 2484297
- [Background] Portenoy RK, Hagen NA. Breakthrough pain: definition, prevalence and characteristics. Pain. 1990 Jun;41(3):273-281. doi: 10.1016/0304-3959(90)90004-W. PMID 1697056
- [Background] Davies AN. Cancer-related breakthrough pain. Br J Hosp Med (Lond). 2006 Aug;67(8):414-6. doi: 10.12968/hmed.2006.67.8.21960. PMID 16918095
- [Background] Greco MT, Corli O, Montanari M, Deandrea S, Zagonel V, Apolone G; Writing Protocol Committee; Cancer Pain Outcome Research Study Group (CPOR SG) Investigators. Epidemiology and pattern of care of breakthrough cancer pain in a longitudinal sample of cancer patients: results from the Cancer Pain Outcome Research Study Group. Clin J Pain. 2011 Jan;27(1):9-18. doi: 10.1097/AJP.0b013e3181edc250. PMID 20842024
- [Background] Deandrea S, Corli O, Consonni D, Villani W, Greco MT, Apolone G. Prevalence of breakthrough cancer pain: a systematic review and a pooled analysis of published literature. J Pain Symptom Manage. 2014 Jan;47(1):57-76. doi: 10.1016/j.jpainsymman.2013.02.015. Epub 2013 Jun 21. PMID 23796584
- See also: Related Info — http://www.marionegri.it/mn/it/index.html